CLINICAL TRIAL: NCT00437333
Title: Insulin Sensitivity After Metformin Suspension in Normal-Weight Women With Polycystic Ovary Syndrome
Brief Title: Metformin Suspension and Insulin Sensitivity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Magna Graecia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MM-187-2004; Prot. 2004063411_003
Record Dates: First submitted 2007-02-20; First posted 2007-02-21 (Estimated); Last update posted 2007-02-21 (Estimated); Status verified 2007-02

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Insulin sensitivity; Insulin-sensitizing drug; Metformin; PCOS; Treatment
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance

INTERVENTIONS:
Drug: Metformin cloridrate

SUMMARY:
Metformin is an insulin sensitizing drug routinely used for the treatment of anovulatory patients with polycystic ovary syndrome (PCOS). To date, the metabolic effects of the long-term metformin administration are know but no data are available on the effects after its suspension.

The purpose of this study is to evaluate the effects of metformin suspension on insulin sensitivity in PCOS patients.

DETAILED DESCRIPTION:
Thirty young normal-weight anovulatory PCOS women will be enrolled. The diagnosis of PCOS will be based on the presence of clinical [Ferriman-Gallwey score ≥ 8] or biochemical hyperandrogenism (serum testosterone levels (>2 SD above our reference mean values) and chronic anovulation [serum luteal progesterone (P) below 2 ng/mL)].

Patients will be randomly allocated into two groups (metformin and placebo group) using a computer-software. Fifteen PCOS patients will be treated with metformin at a dosage of 1700 mg daily (one tablet of 850 mg twice daily; metformin group), whereas other 15 PCOS will be treated with placebo tables (one tablet twice daily; placebo group). The duration of the treatment will be 12 months. Patients will be instructed to follow their usual diet and physical activity, and to use barrier contraception throughout the study. The length and the frequency of the menstrual cycles, and the adverse experiences (AEs) will be reported on a daily diary.

Each subject will undergo follow-up visits under (at six and 12 months from treatment starting) and after treatment (at six and 12 months from treatment withdrawal). At each follow-up visit, in all subjects the same operator will perform clinical, hormonal, metabolic, and insulin sensitivity assessments by euglycemic hyperinsulinemic clamp.

ELIGIBILITY:
Inclusion Criteria:

* Polycystic ovary syndrome (using NIH criteria).

Exclusion Criteria:

* Age <20 or >30 years;
* BMI higher than 25 and lower than 18;
* Neoplastic, metabolic, hepatic, and cardiovascular disorders or other concurrent medical illnesses;
* Hypothyroidism, hyperprolactinemia, Cushing's syndrome, and non-classical congenital adrenal hyperplasia;
* Current or previous use of oral contraceptives, glucocorticoids, antiandrogens, ovulation induction agents, antidiabetic and anti-obesity drugs or other hormonal drugs;
* Intention to start a diet or a specific program of physical activity.

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30
Dates: Start 2003-12; Study Completion 2006-04

PRIMARY OUTCOMES:
Insulin sensitivity by euglycemic hyperinsulinemic clamp

SECONDARY OUTCOMES:
Clinical, hormonal, and metabolic assessments

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Palomba, MD, Principal Investigator — Department of Obstetrics and Gynecology, University "Magna Graecia" of Catanzaro
Locations (1):
- "Pugliese" Hospital, Catanzaro, Italy